CLINICAL TRIAL: NCT01095601
Title: A Phase I, Single-Centre, Open-Label, Randomized, Four-Period Crossover Study to Assess the Effect of Food on the Pharmacokinetics of Avanafil, to Determine The Relative Bioavailability of Two Avanafil Tablet Formulations and to Investigate Dose Proportionality in Healthy Male Subjects
Brief Title: Assess the Effect of Food on Avanafil Pharmacokinetic (PK), to Compare 2 Oral Formulations of Avanafil,and Investigate Dose Proportionality in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Wesley Day, Vivus, Inc
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: TA-020
Record Dates: First submitted 2010-03-28; First posted 2010-03-30 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2011-01

CONDITIONS: Healthy
Keywords: avanafil; absoprion; bioavailability; food effect; dose-proportionality; TA-1790; Pharmacokinetics of avanafil
MeSH Terms: interventions — avanafil

ARMS (4):
- Treatment A (Other): 2x100 mg Formulation II avanafil tablet, fasted
  Interventions: Drug: Avanafil
- Treatment B (Other): 2x100 mg Formulation II avanafil tablet, fed
  Interventions: Drug: Avanafil
- Treatment C (Other): 2x100 mg Formulation I avanafil tablet, fasted
  Interventions: Drug: Avanafil
- Treatment D (Other): 1x50 mg Formulation II avanafil tablet, fasted
  Interventions: Drug: Avanafil

INTERVENTIONS:
Drug: Avanafil — * Treatment A: 2x100 mg Formulation II avanafil tablet, fasted
  * Treatment B: 2x100 mg Formulation II avanafil tablet, fed
  * Treatment C: 2x100 mg Formulation I avanafil tablet, fasted
  * Treatment D: 1x50 mg Formulation II avanafil tablet, fasted
  Other Names: TA-1790

SUMMARY:
This study will assess the effect of food on the pharmacokinetics of avanafil (Formulation II); determine the relative bioavailability of two avanafil tablet formulations (Formulation I versus Formulation II) and will investigate the dose-proportionality of Formulation II avanafil tablet.

DETAILED DESCRIPTION:
In this Phase I, single-centre, open-label, randomized, four-period crossover study, each eligible subject will be randomized to receive the 4 treatments in a 4-way crossover fashion. The 4 treatments are as follows:

* Treatment A: 2x100 mg Formulation II avanafil tablet, fasted
* Treatment B: 2x100 mg Formulation II avanafil tablet, fed
* Treatment C: 2x100 mg Formulation I avanafil tablet, fasted
* Treatment D: 1x50 mg Formulation II avanafil tablet, fasted Subjects will report to the study site on the evening before each treatment and will remain at the site until the 24-hour PK sample has been drawn. A single oral dose of avanafil tablets will be administered with 240 mL of water. A washout period of at least 5 days will occur between the treatments. Subjects in treatment groups A, C and D will fast at least 10 hours prior to and for at least 4 hours following dosing. Subjects in treatment group B will eat a standardized high fat breakfast 30 prior to dosing. Standard meals will be provided uniformly to all subjects at approximately 4 and 9 hours after dosing, and an evening snack will be provided approximately 12 - 13 hours after dosing. Blood samples for the determination of plasma avanafil and its metabolite concentrations will be obtained from each subject at 0 (30 minutes pre-dose), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 8, 12, 18 and 24 hours post-dose in each treatment period.

Adverse events; laboratory evaluations; color vision testing (Treatment A only), electrocardiogram and physical examination, vital signs will be assessed at various times during the study.

ELIGIBILITY:
Inclusion Criteria:

* adult male subjects,
* 18 to 45 years of age,
* must be medically healthy with no clinically significant screening results.

Exclusion Criteria:

* history or clinical evidence of clinically relevant cardiovascular (including thromboembolic disorders), hepatic, renal, hematological, endocrine, pulmonary, gastrointestinal, psychiatric or neurological impairment;
* any clinically significant laboratory abnormalities as judged by the Investigator;
* systolic blood pressure < 90 or >150 mmHg;
* diastolic blood pressure < 50 or > 95 mmHg;
* history of retinitis pigmentosa or nonarteritic anterior ischemic optic neuropathy; allergy to or previous adverse events with PDE5 inhibitors or their constituents;
* use of prescription or over-the-counter drugs that are known to interfere with metabolism by the cytochrome P450 3A4 enzyme within 30 days prior to Day 1 in Period 1;
* use of any investigational drug within 30 days or six half-lives, whichever is longer, prior to Day 1 in Period 1;
* use of any prescription or over-the-counter drugs or herbal remedies within 14 days prior to Day 1 in Period 1;
* history of alcohol or drug abuse within 18 months, history of smoking within 6 months;
* positive urine alcohol test;
* positive cotinine test, positive urine drug screen;
* positive serology for HIV, HCV antibody, HBsAg.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of avanafil | April through May 2010
  Cmax and AUC of avanafil in each period

SECONDARY OUTCOMES:
Safety/AEs of avanafil | April through May, 2010
  Adverse events; laboratory evaluations; color vision testing (Treatment A only), electrocardiogram and physical examination, vital signs will be assessed at various times during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Shiyin Yee, Study Director — VIVUS LLC